CLINICAL TRIAL: NCT05109676
Title: Monitoring of Progesterone Administered in Infertile Patients During a Cycle of Frozen Embryo Transfer: a Population Pharmacokinetic Study.
Brief Title: Monitoring of Progesterone Administered in Infertile Patients During a Cycle of Frozen Embryo Transfer.
Acronym: PEKAPROGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/21/0490
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: IVF
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients having embryo transfert (Experimental): Patients benefit from the usual treatment for frozen embryo transfer with a preparatory cycle of the artificial endometrium: 150 µg of percutaneous estradiol for approximately 11 days and 200 mg of progesterone morning and evening to be taken vaginally for 2 days in case of embryo transfer at day 2 stage, 3 days in case of embryo transfer at day 3 stage, 5 days in case of day 5 embryo transfer or 6 days in case of day 6 embryo transfer.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire will be offered to patients and identify the schedules of administration of progesterone, the day and time of blood samples taken as part of the care, the potential adverse events associated with this administration.

SUMMARY:
During an In Vitro Fertilization (IVF) attempt, several embryos are obtained but not all of them can be transferred to the uterus in the same cycle due to the risk of multiple pregnancies. Thus, it is very common for these couples to benefit from cryopreservation. Patients scheduled for frozen embryo transfer (TEC) receive estrogen and progesterone replacement therapy to prepare the endometrium for implantation. Data from the literature recently showed that low progesterone on the day of embryo transfer was responsible for a significantly higher rate of implantation failure and miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing a frozen embryo transfer in an artificial cycle at the AMP center of the Toulouse University Hospital.
* Affiliation to a social security scheme or equivalent
* Patient fulfilling the conditions for access to the AMP according to French bioethics law
* Patient having given her consent (oral or written) after clear and fair information

Exclusion Criteria:

* Patient who received intramuscular administration of progesterone during the endometrial preparation phase.
* Patient with comprehension difficulties.
* Protected adult patient (safeguard of justice, guardianship or curatorship)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Average plasma progesterone concentration. | Day of embryo transfer.
  Dosage of apparent clearance (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Gatimel, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No